CLINICAL TRIAL: NCT01026818
Title: A Randomised, Double-Blind, Placebo-Controlled Study to Evaluate the Effect on Unassisted Erectile Function of the Early Use of Tadalafil 5 mg Once a Day and Tadalafil 20 mg On Demand Treatment for 9 Months in Subjects Undergoing Bilateral Nerve-Sparing Radical Prostatectomy
Brief Title: A Study of Tadalafil After Radical Prostatectomy
Acronym: REACTT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13086; H6D-EW-LVIK (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Results first posted 2013-11-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2013-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Radical Prostatectomy
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tadalafil daily [5 milligrams (mg)] (Experimental): After the treatment period and 6-week study Drug-Free Period, all participants can continue on study in an optional 5-mg tadalafil 3-month Open-Label Period.
  Interventions: Drug: Tadalafil
- Tadalafil on demand (20 mg) (Experimental): After the treatment period and 6-week study Drug-Free Period, all participants can continue on study in an optional 5-mg tadalafil 3-month Open-Label Period.
  Interventions: Drug: Tadalafil
- Placebo (Placebo Comparator): After the treatment period and 6-week study Drug-Free Period, all participants can continue on study in an optional 5-mg tadalafil 3-month Open-Label Period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil — Administered by mouth for 9 months
  Other Names: Cialis; LY450190
  Arms: Tadalafil daily [5 milligrams (mg)]; Tadalafil on demand (20 mg)
Drug: Placebo — Administered by mouth, daily or on demand for 9 months
  Arms: Placebo

SUMMARY:
The study will include patients with localized prostate cancer who experience erectile dysfunction following bilateral nerve-sparing radical prostatectomy. Patients will be randomly assigned to three treatment arms: Tadalafil 5 mg once a day, Tadalafil 20 mg on demand (prior to anticipated sexual activity), and placebo. Patients will stay on therapy for 9 months and after withdrawal of medication for 6 weeks, patients will be evaluated for recovery of unassisted erectile function (without medication). An open-label extension for three months will evaluate the responsiveness of all patients to Tadalafil 5 mg once a day. Further objectives are to evaluate the treatment satisfaction of the respective therapies.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to undergo Bilateral nerve-sparing radical prostatectomy (BNSRP) for organ-confined, non-metastatic prostate cancer
* have a normal preoperative erectile function score of more or equal to 22 at screening(as evaluated by International Index of Erectile Function - Erectile Function domain (IIEF-EF))
* develop Erectile Dysfunction (ED) (defined as the consistent inability to achieve and/or maintain an erection sufficient to permit satisfactory sexual intercourse) after surgery
* have an interest in resuming sexual activity as soon as possible after surgery and anticipate having the same adult female sexual partner during the study
* agree not to use any other treatment for ED, including herbal and over-the-counter (OTC) medications, during the study
* does not require the initiation of adjuvant therapy for prostate cancer

Exclusion Criteria:

* history of ED
* have received previous or current treatment with tadalafil or any other Phosphodiesterase Type 5 (PDE5) inhibitor
* have undergone, or plan to undergo, radiation or hormonal therapy for prostate cancer
* have a history of prostatic surgery or prostatic physical treatments
* have a history of diabetes mellitus
* have a history of galactose intolerance, lapp lactase deficiency, or glucose-galactose malabsorption
* have clinically significant renal insufficiency as determined by the investigator

Ages: 18 Years to 67 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 583 (Actual)
Dates: Start 2009-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (52):
- Belgium (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kortrijk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
- Canada (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Victoria, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
- France (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Créteil
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grenoble
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nîmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pierre-Bénite
- Germany (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Braunschweig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Herne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leverkusen
- Italy (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Acquavivadellefonti
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergamo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bologna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Perugia
- Netherlands (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., 's-Hertogenbosch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leiden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nijmegen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Veldhoven
- Poland (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bydgoszcz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kielce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zabrze
- Spain (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aravaca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Majadahonda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- Switzerland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Basel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lucerne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zurich
- United Kingdom (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cambridge, Cambridgeshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middlesbrough, Cleveland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stevenage, Herts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Withington, Manchester

REFERENCES:
- [Derived] Montorsi F, Oelke M, Henneges C, Brock G, Salonia A, d'Anzeo G, Rossi A, Mulhall JP, Buttner H. Exploratory Decision-Tree Modeling of Data from the Randomized REACTT Trial of Tadalafil Versus Placebo to Predict Recovery of Erectile Function After Bilateral Nerve-Sparing Radical Prostatectomy. Eur Urol. 2016 Sep;70(3):529-37. doi: 10.1016/j.eururo.2016.02.036. Epub 2016 Mar 3. PMID 26947602
- [Derived] Patel HR, Ilo D, Shah N, Cuzin B, Chadwick D, Andrianne R, Henneges C, Barry J, Hell-Momeni K, Branicka J, Buttner H. Effects of tadalafil treatment after bilateral nerve-sparing radical prostatectomy: quality of life, psychosocial outcomes, and treatment satisfaction results from a randomized, placebo-controlled phase IV study. BMC Urol. 2015 Apr 12;15:31. doi: 10.1186/s12894-015-0022-9. PMID 25879460
- [Derived] Montorsi F, Brock G, Stolzenburg JU, Mulhall J, Moncada I, Patel HR, Chevallier D, Krajka K, Henneges C, Dickson R, Buttner H. Effects of tadalafil treatment on erectile function recovery following bilateral nerve-sparing radical prostatectomy: a randomised placebo-controlled study (REACTT). Eur Urol. 2014 Mar;65(3):587-96. doi: 10.1016/j.eururo.2013.09.051. Epub 2013 Oct 13. PMID 24169081

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of a 6-week screening period including the time of bilateral nerve-sparing radical prostatectomy (BNSRP) surgery, a 9-month, randomized Double-Blind (DB), Placebo-Controlled Treatment Period, followed by a 6-week, Drug-Free Washout Period, and a 3-month, Open-Label (OL) Period.
Groups:
- Screen - BNSRP: BNSRP surgery during Screening Period.
- Tadalafil 5 mg OaD: Tadalafil 5 mg once a day (OaD) + Placebo as required/on demand (PRN) for 9 months during Double-Blind, Placebo-Controlled Treatment Period, followed by a 6-week, Drug-Free Washout Period, and a 3-month, Open-Label Period with tadalafil 5 mg OaD.
- Tadalafil 20 mg PRN: Placebo OaD + Tadalafil 20 mg PRN for 9 months during Double-Blind, Placebo-Controlled Treatment Period, followed by a 6-week, Drug-Free Washout Period, and a 3-month, Open-Label Period with tadalafil 5 mg OaD.
- Placebo: Placebo OaD + Placebo PRN for 9 months during Double-Blind, Placebo-Controlled Treatment Period, followed by a 6-week, Drug-Free Washout Period, and a 3-month, Open-Label Period with tadalafil 5 mg OaD.
Period: Screening Period
Arm/Group | Screen - BNSRP | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Started | 583 | 0 | 0 | 0
Completed | 423 | 0 | 0 | 0
Not Completed | 160 | 0 | 0 | 0
Not completed — Entry Criteria Not Met | 105 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 49 | 0 | 0 | 0
Not completed — Protocol Deviation | 3 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Period: DB Treatment Period (Month 0 - 9)
Arm/Group | Screen - BNSRP | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Started | 0 | 139 | 143 | 141
Received at Least 1 Dose of Study Drug | 0 | 139 | 143 | 141
Completed | 0 | 114 | 122 | 115
Not Completed | 0 | 25 | 21 | 26
Not completed — Adverse Event | 0 | 10 | 6 | 4
Not completed — Withdrawal by Subject | 0 | 7 | 3 | 3
Not completed — Lack of Efficacy | 0 | 3 | 2 | 6
Not completed — Lost to Follow-up | 0 | 3 | 0 | 4
Not completed — Entry Criteria Not Met | 0 | 2 | 9 | 7
Not completed — Protocol Deviation | 0 | 0 | 1 | 2
Period: Drug-Free Washout Period (Month 9-10.5)
Arm/Group | Screen - BNSRP | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Started | 0 | 114 | 122 | 115
Completed | 0 | 105 | 117 | 108
Not Completed | 0 | 9 | 5 | 7
Not completed — Entry Criteria Not Met | 0 | 2 | 1 | 2
Not completed — Lack of Efficacy | 0 | 2 | 1 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 2
Not completed — Physician Decision | 0 | 1 | 1 | 0
Not completed — Sponsor Decision | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0
Not completed — Death | 0 | 0 | 0 | 1
Period: OL Period (Month 10.5 - 13.5)
Arm/Group | Screen - BNSRP | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Started | 0 | 105 | 117 | 108
Completed | 0 | 98 | 112 | 105
Not Completed | 0 | 7 | 5 | 3
Not completed — Entry Criteria Not Met | 0 | 2 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 2 | 1
Not completed — Protocol Deviation | 0 | 1 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo | Total
Number analyzed (Participants) | 139 | 143 | 141 | 423
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (5.07) | 57.5 (5.91) | 57.6 (5.69) | 57.9 (5.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 139 | 143 | 141 | 423
Race/Ethnicity, Customized [Number; unit: participants]
  White | 137 | 141 | 138 | 416
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 1 | 1
  Black or African American | 2 | 1 | 2 | 5
Region of Enrollment [Number; unit: participants]
  France | 12 | 13 | 13 | 38
  Canada | 13 | 13 | 12 | 38
  Belgium | 7 | 9 | 8 | 24
  Poland | 10 | 9 | 8 | 27
  Spain | 38 | 39 | 39 | 116
  Germany | 26 | 25 | 27 | 78
  Netherlands | 0 | 2 | 1 | 3
  United Kingdom | 7 | 8 | 8 | 23
  Switzerland | 1 | 1 | 1 | 3
  Italy | 25 | 24 | 24 | 73

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Score of Greater Than or Equal to 22 in the Erectile Function (EF) Domain of the International Index of Erectile Function (IIEF) Questionnaire
Description: Self-reported erectile function during the past 4 weeks. IIEF- EF is the sum of Questions 1-5 and 15 of the IIEF. Questions 1-5 are scored 0 (no sexual activity for Question 1, no sexual stimulation for Question 2 and did not attempt intercourse for Questions 3-5) to 5 (high erectile function) and Question 15 is scored 1 (very low confidence) to 5 (very high confidence), for a total score ranging from 1 to 30. Higher scores represent better erectile function. Data presented are the percentage of participants with an IIEF-EF Total Score greater than or equal to (≥) 22.
Time Frame: Month 10.5
Population: All randomized participants who received at least 1 dose of study drug and had IIEF-EF Total Scores measurement at Month 10.5.
Measure: Number; unit: percentage of participants
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 139 | 142 | 141
percentage of participants | 20.9 | 16.9 | 19.1
Statistical Analysis 1: Comparison: Tadalafil 5 mg OaD vs Placebo; A sample size of 412 randomized participants provided 84% power to detect a 20% difference in the proportions for the 3 treatment groups. The sample size allowed for a 20% withdrawal during the study; Test type: Superiority or Other; p = 0.675, Regression, Logistic — The Type I error was controlled for multiplicity using a Bonferroni-Hommel procedure. First the largest p-value for the odds ratio to placebo was tested at the 5% level and in case of no rejection the second p-value was tested at the 2.5% level; The logistic regression model included terms for treatment group, country, and age group; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.63 to 2.06]
Statistical Analysis 2: Comparison: Tadalafil 20 mg PRN vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.704, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; The logistic regression model included terms for treatment group, country, and age group; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.48 to 1.65]

2. Secondary Outcome: Percentage of Participants With a Score of Greater Than or Equal to 22 in the International Index of Erectile Function- Erectile Function (IIEF-EF) Domain
Description: as for outcome 1
Time Frame: Month 9 and Month 13.5
Population: All randomized participants who received at least 1 dose of study drug and had IIEF-EF Total Scores measurements at Months 9 and 13.5.
Measure: Number; unit: percentage of participants
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 139 | 142 | 141
percentage of participants
  Month 9 | 25.2 | 19.7 | 14.2
  Month 13.5 | 32.4 | 33.1 | 27.0
Statistical Analysis 1: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.016, Regression, Logistic — P-value is for Month 9; The logistic regression model included terms for treatment group, country, and age group; Odds Ratio (OR) = 2.15, 95% CI 2-sided [1.16 to 3.99]
Statistical Analysis 2: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.210, Regression, Logistic — P-value is for Month 9; The logistic regression model included terms for treatment group, country, and age group; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.79 to 2.85]
Statistical Analysis 3: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.273, Regression, Logistic — P-value is for Month 13.5; The logistic regression model included terms for treatment group, country, and age group; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.79 to 2.28]
Statistical Analysis 4: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.259, Regression, Logistic — P-value is for Month 13.5; The logistic regression model included terms for treatment group, country, and age group; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.80 to 2.29]

3. Secondary Outcome: Change From Baseline to Endpoint in the International Index of Erectile Function- Erectile Function (IIEF-EF) Total Score
Description: Self-reported erectile function during the past 4 weeks. IIEF- EF is the sum of Questions 1-5 and 15 of the IIEF. Questions 1-5 are scored 0 (no sexual activity for Question 1, no sexual stimulation for Question 2 and did not attempt intercourse for Questions 3-5) to 5 (high erectile function) and Question 15 is scored 1 (very low confidence) to 5 (very high confidence), for a total score ranging from 1 to 30. Higher scores represent better erectile function. The Mixed Model for Repeated Measures (MMRM) analysis was used to calculate Least Squares (LS) mean and 95% confidence interval (CI). LS mean values are adjusted for baseline score, treatment, country, visit, visit-by-treatment, age group, and age group-by-treatment (if significant at p<0.10).
Time Frame: Randomization (Baseline), Months 9 and 10.5 and 13.5
Population: All randomized participants who received at least 1 dose of study drug, had baseline and at least one post-baseline IIEF-EF Total Scores measurement at Months 9, 10.5 and 13.5.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 139 | 142 | 141
units on a scale
  Month 9 | 7.73 [5.73 to 9.73] | 6.53 [4.56 to 8.50] | 4.93 [2.88 to 6.98]
  Month 10.5 | 6.24 [4.22 to 8.25] | 5.76 [3.78 to 7.73] | 5.98 [3.92 to 8.03]
  Month 13.5 | 10.60 [8.39 to 12.80] | 9.78 [7.63 to 11.92] | 8.97 [6.74 to 11.21]
Statistical Analysis 1: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis — P-value is for Month 9; The MMRM model included baseline, treatment, country, visit, visit-by-treatment, age group, and age group-by-treatment (if significant at p<0.10); LS Mean Differences = 2.80, 95% CI 2-sided [0.76 to 4.83], Standard Error of Mean 1.03
Statistical Analysis 2: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.118, Mixed Models Analysis — P-value is for Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean differences = 1.59, 95% CI 2-sided [-0.41 to 3.60], Standard Error of Mean 1.02
Statistical Analysis 3: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.802, Mixed Models Analysis — P-value is for Month 10.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.26, 95% CI 2-sided [-1.79 to 2.31], Standard Error of Mean 1.04
Statistical Analysis 4: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.830, Mixed Models Analysis — P-value is for Month 10.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = -0.22, 95% CI 2-sided [-2.23 to 1.79], Standard Error of Mean 1.02
Statistical Analysis 5: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.184, Mixed Models Analysis — P-value is for Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 1.62, 95% CI 2-sided [-0.78 to 4.03], Standard Error of Mean 1.22
Statistical Analysis 6: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.500, Mixed Models Analysis — P-value is for Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.81, 95% CI 2-sided [-1.54 to 3.16], Standard Error of Mean 1.20

4. Secondary Outcome: Change From Baseline to Endpoint in the International Index of Erectile Function (IIEF) Domains (Intercourse Satisfaction Domain, Orgasmic Function Domain, Sexual Desire Domain, Overall Satisfaction Domain)
Description: Self-reported overall satisfaction during past 4 weeks. Orgasmic function score is sum of Questions (Q)9 and 10 of IIEF. Scores range from 0 (no sexual stimulation or intercourse) to 5 (high orgasm) for each Q, total 0 to 10. Sexual desire score is sum of Q11 and 12 of IIEF. Scores range from 1 (low/no desire) to 5 (high desire) for each Q, total 2 to 10. Intercourse satisfaction score is sum of Q6, 7 and 8 of IIEF. Scores range from 0 (no attempts for Q6, did not attempt intercourse for Q7 and no intercourse for Q8) to 5 (high satisfaction) for each Q, total 0 to 15. Overall satisfaction score is sum of Q13 and 14 of IIEF. Scores range from 1 (low/no satisfaction) to 5 (high satisfaction) for each Q, total 2 to 10. Higher total scores for each domain indicate higher function. MMRM analysis was used to calculate LS mean and 95% CI. LS mean values are adjusted for baseline, treatment, country, visit, visit-by-treatment, age group, and age group-by-treatment (if significant at p<0.10).
Time Frame: Randomization (Baseline), Months 9 and 10.5 and 13.5
Population: All randomized participants who received at least 1 dose of study drug, had baseline and at least one post-baseline IIEF domain scores measurements at Months 9, 10.5 and 13.5.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 139 | 142 | 141
units on a scale
  Orgasmic function - Month 9 | 2.76 [1.98 to 3.55] | 2.48 [1.70 to 3.26] | 2.39 [1.59 to 3.19]
  Orgasmic function - Month 10.5 | 2.94 [2.13 to 3.76] | 2.48 [1.68 to 3.28] | 2.48 [1.66 to 3.31]
  Orgasmic function - Month 13.5 | 3.57 [2.75 to 4.39] | 2.90 [2.10 to 3.70] | 3.42 [2.59 to 4.25]
  Sexual desire - Month 9 | 0.65 [0.18 to 1.12] | 0.65 [0.18 to 1.11] | 0.63 [0.15 to 1.11]
  Sexual desire - Month 10.5 | 0.61 [0.14 to 1.07] | 0.65 [0.20 to 1.11] | 0.55 [0.08 to 1.01]
  Sexual desire - Month 13.5 | 1.04 [0.56 to 1.52] | 0.89 [0.42 to 1.35] | 0.95 [0.46 to 1.43]
  Intercourse satisfaction - Month 9 | 3.89 [2.90 to 4.88] | 3.50 [2.52 to 4.48] | 2.96 [1.95 to 3.96]
  Intercourse satisfaction - Month 10.5 | 3.21 [2.19 to 4.22] | 2.81 [1.81 to 3.81] | 2.72 [1.69 to 3.75]
  Intercourse satisfaction - Month 13.5 | 4.70 [3.65 to 5.75] | 4.08 [3.05 to 5.10] | 4.14 [3.08 to 5.20]
  Overall satisfaction - Month 9 | 0.97 [0.38 to 1.56] | 0.93 [0.35 to 1.51] | 0.78 [0.18 to 1.38]
  Overall satisfaction - Month 10.5 | 0.64 [0.05 to 1.23] | 0.48 [-0.10 to 1.06] | 0.72 [0.12 to 1.32]
  Overall satisfaction - Month 13.5 | 1.50 [0.87 to 2.13] | 1.57 [0.96 to 2.19] | 1.52 [0.88 to 2.15]
Statistical Analysis 1: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.340, Mixed Models Analysis — P-value is for orgasmic function - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.37, 95% CI [-0.39 to 1.14], Standard Error of Mean 0.39
Statistical Analysis 2: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.821, Mixed Models Analysis — P-value is for orgasmic function - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.09, 95% CI 2-sided [-0.67 to 0.84], Standard Error of Mean 0.38
Statistical Analysis 3: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.268, Mixed Models Analysis — P-value is for orgasmic function - Month 10.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.46, 95% CI 2-sided [-0.36 to 1.28], Standard Error of Mean 0.42
Statistical Analysis 4: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.998, Mixed Models Analysis — P-value is for orgasmic function - Month 10.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = -0.00, 95% CI 2-sided [-0.80 to 0.80], Standard Error of Mean 0.41
Statistical Analysis 5: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.728, Mixed Models Analysis — P-value is for orgasmic function - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.15, 95% CI 2-sided [-0.68 to 0.97], Standard Error of Mean 0.42
Statistical Analysis 6: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.203, Mixed Models Analysis — P-value is for orgasmic function - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = -0.52, 95% CI 2-sided [-1.33 to 0.28], Standard Error of Mean 0.41
Statistical Analysis 7: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.950, Mixed Models Analysis — P-value is for sexual desire - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.02, 95% CI 2-sided [-0.46 to 0.49], Standard Error of Mean 0.24
Statistical Analysis 8: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.950, Mixed Models Analysis — P-value is for sexual desire - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.01, 95% CI 2-sided [-0.45 to 0.48], Standard Error of Mean 0.24
Statistical Analysis 9: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.792, Mixed Models Analysis — P-value is for sexual desire - Month 10.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.06, 95% CI 2-sided [-0.39 to 0.51], Standard Error of Mean 0.23
Statistical Analysis 10: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.631, Mixed Models Analysis — P-value is for sexual desire - Month 10.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.11, 95% CI 2-sided [-0.34 to 0.55], Standard Error of Mean 0.23
Statistical Analysis 11: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.691, Mixed Models Analysis — P-value is for sexual desire - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.10, 95% CI 2-sided [-0.38 to 0.58], Standard Error of Mean 0.24
Statistical Analysis 12: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.801, Mixed Models Analysis — P-value is for sexual desire - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = -0.06, 95% CI 2-sided [-0.53 to 0.41], Standard Error of Mean 0.24
Statistical Analysis 13: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.065, Mixed Models Analysis — P-value is for intercourse satisfaction - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.93, 95% CI 2-sided [-0.06 to 1.92], Standard Error of Mean 0.50
Statistical Analysis 14: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.274, Mixed Models Analysis — P-value is for intercourse satisfaction - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.54, 95% CI 2-sided [-0.43 to 1.51], Standard Error of Mean 0.49
Statistical Analysis 15: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.359, Mixed Models Analysis — P-value is for intercourse satisfaction - Month 10.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.48, 95% CI 2-sided [-0.55 to 1.52], Standard Error of Mean 0.53
Statistical Analysis 16: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.863, Mixed Models Analysis — P-value is for intercourse satisfaction - Month 10.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.09, 95% CI 2-sided [-0.93 to 1.11], Standard Error of Mean 0.52
Statistical Analysis 17: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.314, Mixed Models Analysis — P-value is for intercourse satisfaction - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.56, 95% CI 2-sided [-0.53 to 1.66], Standard Error of Mean 0.56
Statistical Analysis 18: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.910, Mixed Models Analysis — P-value is for intercourse satisfaction - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = -0.06, 95% CI 2-sided [-1.13 to 1.01], Standard Error of Mean 0.54
Statistical Analysis 19: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.532, Mixed Models Analysis — P-value is for overall satisfaction - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.19, 95% CI 2-sided [-0.40 to 0.78], Standard Error of Mean 0.30
Statistical Analysis 20: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.620, Mixed Models Analysis — P-value is for overall satisfaction - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.15, 95% CI 2-sided [-0.43 to 0.73], Standard Error of Mean 0.30
Statistical Analysis 21: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.792, Mixed Models Analysis — P-value is for overall satisfaction - Month 10.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = -0.08, 95% CI 2-sided [-0.67 to 0.51], Standard Error of Mean 0.30
Statistical Analysis 22: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.410, Mixed Models Analysis — P-value is for overall satisfaction - Month 10.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = -0.24, 95% CI 2-sided [-0.82 to 0.34], Standard Error of Mean 0.29
Statistical Analysis 23: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.955, Mixed Models Analysis — P-value is for overall satisfaction - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = -0.02, 95% CI [-0.68 to 0.65], Standard Error of Mean 0.34
Statistical Analysis 24: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.868, Mixed Models Analysis — P-value is for overall satisfaction - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.05, 95% CI 2-sided [-0.59 to 0.70], Standard Error of Mean 0.33

5. Secondary Outcome: Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) Questionnaire Mean Score
Description: The EDITS questionnaire is a validated questionnaire consisting of 11 questions evaluating self-reported satisfaction with the erectile dysfunction (ED) treatment. Responses were based on the experiences during the previous 4 weeks. Each question is rated on a scale of 0 (extremely low treatment satisfaction) to 4 (extremely high treatment satisfaction). The EDITS mean score was obtained by adding each individual result for all questions, dividing by the number of questions answered. The mean scores range from 0 (extremely low treatment satisfaction) to 4 (extremely high satisfaction). The Mixed Model for Repeated Measures (MMRM) analysis was used to calculate Least Squares (LS) mean and 95% Confidence Interval (CI). LS mean values are adjusted for treatment, country, visit, visit-by-treatment, age group, and age group-by-treatment (if significant at p<0.10).
Time Frame: Months 9 and 13.5
Population: All randomized participants who received at least 1 dose of study drug and had EDITS mean scores measurements at Months 9 and 13.5.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 139 | 142 | 141
units on a scale
  Month 9 | 2.21 (0.11) [2.00 to 2.42] | 2.11 [1.92 to 2.30] | 1.88 [1.67 to 2.09]
  Month 13.5 | 2.54 [2.31 to 2.77] | 2.38 [2.17 to 2.59] | 2.25 [2.03 to 2.48]
Statistical Analysis 1: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis — P-value is for Month 9; The MMRM model included terms for treatment, country, visit, visit-by-treatment, age group, and age group-by-treatment (if significant at p<0.10); LS Mean Differences = 0.33, 95% CI 2-sided [0.10 to 0.56], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.041, Mixed Models Analysis — P-value is for Month 9; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 0.23, 95% CI 2-sided [0.01 to 0.45], Standard Error of Mean 0.11
Statistical Analysis 3: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.035, Mixed Models Analysis — P-value is for Month 13.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 0.28, 95% CI [0.02 to 0.54], Standard Error of Mean 0.13
Statistical Analysis 4: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.316, Mixed Models Analysis — P-value is for Month 13.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 0.13, 95% CI 2-sided [-0.12 to 0.38], Standard Error of Mean 0.13

6. Secondary Outcome: Change From Baseline in Self Esteem and Relationship (SEAR) Questionnaire Score
Description: The SEAR questionnaire is a participant-reported measure of psychosocial outcomes in men with erectile dysfunction (ED). It consists of 14 items. Sexual Relationship domain consists of 8 items (items 1-8). Items 2-8 are rated on a scale of 1 (Never) to 5 (Always), whereas item 1 is reverse scored (1=Always and 5=Never). The total scores for sexual relationship domain range from 8-40 with higher scores indicating better relationship. Self-Esteem subdomain contains items 9 through 12 rated on a scale of 1 (no/low self-esteem) to 5 (high self-esteem). Total scores for Self-Esteem subscale range from 4-20 with higher scores indicating higher self-esteem. The Mixed Model for Repeated Measures (MMRM) analysis was used to calculate Least Squares (LS) mean and 95% Confidence Interval (CI). LS mean values are adjusted for baseline domain score, treatment, country, visit, visit-by-treatment, age group, and age group-by-treatment (if significant at p<0.10).
Time Frame: Randomization (Baseline), Months 9 and 13.5
Population: All randomized participants who received at least 1 dose of study drug, had baseline and at least 1 post-baseline SEAR scores measurement at Months 9 and 13.5.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 139 | 142 | 141
units on a scale
  Sexual relationship - Month 9 | 4.78 [2.87 to 6.68] | 3.50 [1.61 to 5.38] | 3.02 [1.09 to 4.95]
  Sexual relationship - Month 13.5 | 6.90 [4.79 to 9.00] | 6.68 [4.62 to 8.74] | 6.72 [4.62 to 8.83]
  Self-esteem - Month 9 | 0.78 [-0.31 to 1.87] | 0.79 [-0.29 to 1.87] | 0.51 [-0.61 to 1.62]
  Self-esteem - Month 13.5 | 1.67 [0.54 to 2.81] | 1.72 [0.61 to 2.83] | 1.62 [0.47 to 2.77]
Statistical Analysis 1: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.086, Mixed Models Analysis — P-value is for sexual relationship - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 1.75, 95% CI 2-sided [-0.25 to 3.76], Standard Error of Mean 1.02
Statistical Analysis 2: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.637, Mixed Models Analysis — P-value is for sexual relationship - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.47, 95% CI 2-sided [-1.50 to 2.45], Standard Error of Mean 1.00
Statistical Analysis 3: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.885, Mixed Models Analysis — P-value is for sexual relationship - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.17, 95% CI 2-sided [-2.18 to 2.53], Standard Error of Mean 1.20
Statistical Analysis 4: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.972, Mixed Models Analysis — P-value is for sexual relationship - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = -0.04, 95% CI 2-sided [-2.34 to 2.25], Standard Error of Mean 1.17
Statistical Analysis 5: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.621, Mixed Models Analysis — P-value is for self-esteem - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.27, 95% CI 2-sided [-0.81 to 1.36], Standard Error of Mean 0.55
Statistical Analysis 6: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.598, Mixed Models Analysis — P-value is for self-esteem - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.29, 95% CI 2-sided [-0.78 to 1.35], Standard Error of Mean 0.54
Statistical Analysis 7: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.923, Mixed Models Analysis — P-value is for self-esteem - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.06, 95% CI 2-sided [-1.10 to 1.21], Standard Error of Mean 0.59
Statistical Analysis 8: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.857, Mixed Models Analysis — P-value is for self-esteem - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.10, 95% CI 2-sided [-1.03 to 1.24], Standard Error of Mean 0.58

7. Secondary Outcome: Global Assessment Questions (GAQ) Question 1 at Month 9
Description: GAQ Question 1: Choose the one number which best describes how you perceive your ability to achieve and maintain your erections now, compared to how it was before you began taking medication in this study. Responses range from very much better (1) to very much worse (7).
Time Frame: Month 9
Population: All randomized participants who received at least 1 dose of study drug and had GAQ Q1 assessed at Month 9.
Measure: Number; unit: participants
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 114 | 122 | 115
participants
  Very much better | 9 | 10 | 4
  Much better | 12 | 22 | 9
  A little better | 33 | 32 | 22
  No change | 31 | 28 | 48
  A little worse | 4 | 5 | 3
  Much worse | 6 | 8 | 6
  Very much worse | 8 | 11 | 14
  Missing | 11 | 6 | 9

8. Secondary Outcome: Global Assessment Question (GAQ) Question 1 at Month 13.5
Description: as for outcome 7
Time Frame: Month 13.5
Population: All randomized participants who received at least 1 dose of study drug and had GAQ Q1 assessed at Month 13.5.
Measure: Number; unit: participants
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 100 | 114 | 106
participants
  Very much better | 13 | 19 | 16
  Much better | 24 | 25 | 18
  A little Better | 28 | 27 | 28
  No Change | 19 | 23 | 26
  A little worse | 4 | 4 | 2
  Much worse | 3 | 3 | 5
  Very much worse | 5 | 6 | 6
  Missing | 4 | 7 | 5

9. Secondary Outcome: Global Assessment Question (GAQ) Question 2 at Month 9
Description: GAQ Question 2: Choose the one number which best describes how you perceive your sexual life is now, compared to how it was before you began taking medication in this study. Responses range from very much better (1) to very much worse (7).
Time Frame: Month 9
Population: All randomized participants who received at least 1 dose of study drug and had GAQ Q2 assessed at Month 9.
Measure: Number; unit: participants
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 114 | 122 | 115
participants
  Very much better | 7 | 7 | 3
  Much better | 12 | 25 | 11
  A little better | 30 | 26 | 18
  No change | 31 | 27 | 49
  A little worse | 8 | 10 | 4
  Much worse | 7 | 10 | 10
  Very much worse | 9 | 9 | 11
  Missing | 10 | 8 | 9

10. Secondary Outcome: Global Assessment Question (GAQ) Question 2 at Month 13.5
Description: as for outcome 9
Time Frame: Month 13.5
Population: All randomized participants who received at least 1 dose of study drug and had GAQ Q2 assessed at Month 13.5.
Measure: Number; unit: participants
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 100 | 114 | 106
participants
  Very much better | 9 | 20 | 14
  Much better | 29 | 23 | 21
  A little better | 20 | 26 | 24
  No change | 25 | 24 | 26
  A little worse | 4 | 5 | 5
  Much worse | 4 | 3 | 7
  Very much worse | 5 | 6 | 4
  Missing | 4 | 7 | 5

11. Secondary Outcome: Residual Erectile Function (REF) at Baseline
Description: The participant is asked to rate the hardness of his erection using a 5-point grading system, with 0 (penis does not enlarge), 1 (penis is larger but not hard), 2 (penis is hard but not enough for penetration), 3 (penis is hard enough for penetration but not completely hard), 4 (penis is completely hard and fully rigid.)
Time Frame: Baseline
Population: All randomized participants who received at least 1 dose of study drug and had REF assessed at baseline.
Measure: Number; unit: participants
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 139 | 142 | 141
participants
  REF = 0 | 61 | 62 | 64
  REF = 1 | 46 | 48 | 47
  REF = 2 | 18 | 17 | 17
  REF = 3 | 12 | 11 | 13
  REF = 4 | 0 | 2 | 0
  Missing | 2 | 2 | 0

12. Secondary Outcome: Residual Erectile Function (REF) at Month 2
Description: as for outcome 11
Time Frame: Month 2
Population: All randomized participants who received at least 1 dose of study drug and had REF assessed at Month 2.
Measure: Number; unit: participants
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 139 | 142 | 141
participants
  REF = 0 | 28 | 27 | 38
  REF = 1 | 38 | 51 | 53
  REF = 2 | 26 | 28 | 19
  REF = 3 | 25 | 23 | 15
  REF = 4 | 9 | 5 | 5
  Missing | 13 | 8 | 11

13. Secondary Outcome: Residual Erectile Function (REF) at Month 5
Description: as for outcome 11
Time Frame: Month 5
Population: All randomized participants who received at least 1 dose of study drug and had REF assessed at Month 5.
Measure: Number; unit: participants
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 123 | 128 | 123
participants
  REF = 0 | 12 | 21 | 27
  REF = 1 | 37 | 39 | 35
  REF = 2 | 19 | 21 | 27
  REF = 3 | 32 | 34 | 19
  REF = 4 | 15 | 6 | 6
  Missing | 8 | 7 | 9

14. Secondary Outcome: Residual Erectile Function (REF) at Month 9
Description: as for outcome 11
Time Frame: Month 9
Population: All randomized participants who received at least 1 dose of study drug and had REF assessed at Month 9.
Measure: Number; unit: participants
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 114 | 122 | 115
participants
  REF = 0 | 11 | 17 | 23
  REF = 1 | 25 | 28 | 35
  REF = 2 | 22 | 30 | 23
  REF = 3 | 23 | 27 | 18
  REF = 4 | 20 | 15 | 10
  Missing | 13 | 5 | 6

15. Secondary Outcome: Residual Erectile Function (REF) at Month 10.5
Description: as for outcome 11
Time Frame: Month 10.5
Population: All randomized participants who received at least 1 dose of study drug and had REF assessed at Month 10.5.
Measure: Number; unit: participants
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 105 | 117 | 108
participants
  REF = 0 | 13 | 17 | 22
  REF = 1 | 29 | 30 | 29
  REF = 2 | 25 | 23 | 19
  REF = 3 | 22 | 31 | 22
  REF = 4 | 12 | 10 | 14
  Missing | 4 | 6 | 2

16. Secondary Outcome: Residual Erectile Function (REF) at Month 13.5
Description: as for outcome 11
Time Frame: Month 13.5
Population: All randomized participants who received at least 1 dose of study drug and had REF assessed at Month 13.5.
Measure: Number; unit: participants
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 100 | 114 | 106
participants
  REF = 0 | 5 | 8 | 11
  REF = 1 | 19 | 20 | 25
  REF = 2 | 17 | 20 | 15
  REF = 3 | 34 | 34 | 28
  REF = 4 | 21 | 28 | 24
  Missing | 4 | 4 | 3

17. Secondary Outcome: Change From Baseline in 'Yes' Answers to Questions 1 to 5 of the Sexual Encounter Profile (SEP)
Description: Participant-assessed diary has 5 questions: Question (Q)1: erection achievement, Q2: successful penetration, Q3: successful intercourse, Q4: satisfied with erection, and Q5: satisfied with sexual experience) for each sexual encounter made over a specified period of time. SEP Q1-Q5 scores were determined as the percentage of 'Yes' responses to each of the 5 questions out of all sexual attempts recorded during the time period. The Mixed Model for Repeated Measures (MMRM) analysis was used to calculate Least Squares (LS) mean and 95% confidence interval (CI). LS mean values are adjusted for treatment, country, visit, visit-by-treatment, age group, and age group-by-treatment (if significant at p<0.10).
Time Frame: Randomization (Baseline), Months 9 and 10.5 and 13.5
Population: All randomized participants who received at least 1 dose of study drug, had baseline and at least 1 post-baseline SEP questions answered at Months 9, 10.5 and 13.5.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of "yes" responses
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 139 | 142 | 141
percentage of "yes" responses
  Q1 - Month 9 | 67.41 [58.29 to 76.54] | 63.88 [55.32 to 72.44] | 52.54 [43.62 to 61.46]
  Q1 - Month 10.5 | 67.78 [58.05 to 77.50] | 64.24 [55.06 to 73.41] | 58.86 [49.15 to 68.58]
  Q1 - Month 13.5 | 86.16 [77.82 to 94.51] | 79.79 [71.93 to 87.65] | 75.27 [66.93 to 83.60]
  Q2 - Month 9 | 44.00 [35.22 to 52.78] | 34.29 [26.03 to 42.56] | 27.67 [19.11 to 36.23]
  Q2 - Month 10.5 | 40.81 [31.21 to 50.40] | 34.99 [25.91 to 44.08] | 36.26 [26.67 to 45.85]
  Q2 - Month 13.5 | 63.48 [53.87 to 73.09] | 56.07 [46.91 to 65.24] | 50.11 [40.56 to 59.67]
  Q3 - Month 9 | 33.67 [25.47 to 41.86] | 24.09 [16.36 to 31.82] | 21.61 [13.62 to 29.59]
  Q3 - Month 10.5 | 28.75 [19.92 to 37.57] | 23.01 [14.65 to 31.37] | 28.52 [19.68 to 37.36]
  Q3 - Month 13.5 | 52.41 [42.80 to 62.02] | 45.83 [36.63 to 55.04] | 40.75 [31.18 to 50.31]
  Q4 - Month 9 | 26.17 [18.93 to 33.40] | 18.15 [11.31 to 24.99] | 14.30 [7.25 to 21.35]
  Q4 - Month 10.5 | 16.94 [9.66 to 24.23] | 11.74 [4.84 to 18.64] | 18.88 [11.54 to 26.22]
  Q4 - Month 13.5 | 42.08 [32.99 to 51.18] | 35.62 [26.88 to 44.37] | 30.56 [21.48 to 39.65]
  Q5 - Month 9 | 25.42 [18.29 to 32.55] | 17.73 [10.99 to 24.47] | 14.04 [7.09 to 20.99]
  Q5 - Month 10.5 | 16.26 [9.21 to 23.31] | 10.52 [3.85 to 17.19] | 19.11 [12.00 to 26.23]
  Q5 - Month 13.5 | 40.81 [31.82 to 49.81] | 34.96 [26.31 to 43.62] | 29.38 [20.39 to 38.37]
Statistical Analysis 1: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis — P-value is for Q1 - Month 9; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 14.87, 95% CI 2-sided [3.92 to 25.83], Standard Error of Mean 5.57
Statistical Analysis 2: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.038, Mixed Models Analysis — P-value is for Q1 - Month 9; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 11.34, 95% CI 2-sided [0.63 to 22.04], Standard Error of Mean 5.45
Statistical Analysis 3: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.148, Mixed Models Analysis — P-value is for Q1 - Month 10.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 8.91, 95% CI 2-sided [-3.18 to 21.00], Standard Error of Mean 6.15
Statistical Analysis 4: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.373, Mixed Models Analysis — P-value is for Q1 - Month 10.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 5.37, 95% CI 2-sided [-6.48 to 17.23], Standard Error of Mean 6.03
Statistical Analysis 5: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.029, Mixed Models Analysis — P-value is for Q1 - Month 13.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 10.90, 95% CI 2-sided [1.14 to 20.66], Standard Error of Mean 4.96
Statistical Analysis 6: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.357, Mixed Models Analysis — P-value is for Q1 - Month 13.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 4.53, 95% CI 2-sided [-5.12 to 14.17], Standard Error of Mean 4.91
Statistical Analysis 7: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — P-value is for Q2 - Month 9; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 16.33, 95% CI 2-sided [5.68 to 26.98], Standard Error of Mean 5.42
Statistical Analysis 8: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.212, Mixed Models Analysis — P-value is for Q2 - Month 9; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 6.62, 95% CI 2-sided [-3.80 to 17.04], Standard Error of Mean 5.30
Statistical Analysis 9: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.461, Mixed Models Analysis — P-value is for Q2 - Month 10.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 4.55, 95% CI 2-sided [-7.58 to 16.68], Standard Error of Mean 6.17
Statistical Analysis 10: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.835, Mixed Models Analysis — P-value is for Q2 - Month 10.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = -1.26, 95% CI 2-sided [-13.16 to 10.63], Standard Error of Mean 6.05
Statistical Analysis 11: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.030, Mixed Models Analysis — P-value is for Q2 - Month13.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 13.36, 95% CI 2-sided [1.27 to 25.46], Standard Error of Mean 6.15
Statistical Analysis 12: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.326, Mixed Models Analysis — P-value is for Q2 - Month13.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 5.96, 95% CI 2-sided [-5.97 to 17.89], Standard Error of Mean 6.07
Statistical Analysis 13: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.019, Mixed Models Analysis — P-value is for Q3 - Month 9; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 12.06, 95% CI [1.98 to 22.15], Standard Error of Mean 5.13
Statistical Analysis 14: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.621, Mixed Models Analysis — P-value is for Q3 - Month 9; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 2.48, 95% CI 2-sided [-7.38 to 12.35], Standard Error of Mean 5.02
Statistical Analysis 15: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.968, Mixed Models Analysis — P-value is for Q3 - Month 10.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 0.23, 95% CI [-11.03 to 11.49], Standard Error of Mean 5.73
Statistical Analysis 16: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.327, Mixed Models Analysis — P-value is for Q3 - Month 10.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = -5.51, 95% CI 2-sided [-16.55 to 5.54], Standard Error of Mean 5.62
Statistical Analysis 17: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.066, Mixed Models Analysis — P-value is for Q3 - Month 13.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 11.67, 95% CI 2-sided [-0.76 to 24.09], Standard Error of Mean 6.32
Statistical Analysis 18: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.415, Mixed Models Analysis — P-value is for Q3 - Month 13.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 5.09, 95% CI 2-sided [-7.17 to 17.34], Standard Error of Mean 6.23
Statistical Analysis 19: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis — P-value is for Q4 - Month 9; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 11.87, 95% CI 2-sided [2.79 to 20.94], Standard Error of Mean 4.61
Statistical Analysis 20: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.394, Mixed Models Analysis — P-value is for Q4 - Month 9; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 3.85, 95% CI 2-sided [-5.03 to 12.72], Standard Error of Mean 4.51
Statistical Analysis 21: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.684, Mixed Models Analysis — P-value is for Q4 - Month 10.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = -1.94, 95% CI 2-sided [-11.28 to 7.41], Standard Error of Mean 4.75
Statistical Analysis 22: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.126, Mixed Models Analysis — P-value is for Q4 - Month 10.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = -7.14, 95% CI 2-sided [-16.30 to 2.02], Standard Error of Mean 4.66
Statistical Analysis 23: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.061, Mixed Models Analysis — P-value is for Q4 - Month 13.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 11.52, 95% CI 2-sided [-0.53 to 23.57], Standard Error of Mean 6.13
Statistical Analysis 24: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.403, Mixed Models Analysis — P-value is for Q4 - Month13.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 5.06, 95% CI 2-sided [-6.83 to 16.95], Standard Error of Mean 6.05
Statistical Analysis 25: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis — P-value is for Q5 - Month 9; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 11.38, 95% CI [2.38 to 20.38], Standard Error of Mean 4.58
Statistical Analysis 26: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.410, Mixed Models Analysis — P-value is for Q5 - Month 9; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 3.69, 95% CI 2-sided [-5.11 to 12.49], Standard Error of Mean 4.47
Statistical Analysis 27: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.537, Mixed Models Analysis — P-value is for Q5 - Month 10.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = -2.85, 95% CI 2-sided [-11.92 to 6.22], Standard Error of Mean 4.61
Statistical Analysis 28: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.058, Mixed Models Analysis — P-value is for Q5 - Month 10.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = -8.59, 95% CI 2-sided [-17.48 to 0.30], Standard Error of Mean 4.52
Statistical Analysis 29: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.061, Mixed Models Analysis — P-value is for Q5 - Month 13.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 11.44, 95% CI 2-sided [-0.54 to 23.41], Standard Error of Mean 6.09
Statistical Analysis 30: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.353, Mixed Models Analysis — P-value is for Q5 - Month 13.5; [statistical method as in outcome 5, analysis 1]; LS Mean Differences = 5.59, 95% CI 2-sided [-6.23 to 17.40], Standard Error of Mean 6.01

18. Secondary Outcome: Change From Baseline in 'Yes' Answers to Morning Erections
Description: The participants were asked to complete the morning erections diary every morning during the 4-week period before randomization and during the 6-week, Drug-Free, Washout Period. Data presented are the changes in the participant's percentage of "yes" responses relative to the number of days the question was answered during treatment. The analysis of covariance (ANCOVA) was used to calculate Least Square (LS) mean and 95% confidence interval (CI). LS mean values are adjusted for treatment, baseline morning erections frequency, age group and country.
Time Frame: Randomization (Baseline), Month 10.5
Population: All randomized participants who received at least 1 dose of study drug and had morning erection question answered at Baseline and Month 10.5.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of "yes" response
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 139 | 142 | 141
percentage of "yes" response | 8.92 [1.45 to 16.39] | 12.16 [5.16 to 19.16] | 14.04 [6.74 to 21.35]
Statistical Analysis 1: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.162, ANCOVA; ANCOVA model included treatment, baseline, age group, and country; LS Mean Differences = -5.12, 95% CI 2-sided [-12.32 to 2.08], Standard Error of Mean 3.66
Statistical Analysis 2: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.603, ANCOVA; ANCOVA model included treatment, baseline, age group, and country; LS Mean Differences = -1.88, 95% CI [-8.99 to 5.24], Standard Error of Mean 3.61

19. Secondary Outcome: Standardized Morning Erections Question (SMEQ) Score at Month 2
Description: Participants evaluated the frequency of their morning erections during the past 3-month period by answering the SMEQ ("Do you ever wake up with an erection") using a 4-point grading system ranging from 0 (Yes, regularly) to 3 (never).
Time Frame: Month 2
Population: All randomized participants who received at least 1 dose of study drug and had SMEQ measurement at Month 2
Measure: Number; unit: participants
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 139 | 142 | 141
participants
  Yes, regularly | 4 | 7 | 7
  Less frequently than in the past | 8 | 15 | 10
  Only occasionally | 41 | 31 | 26
  Never | 73 | 80 | 87
  Missing | 13 | 9 | 11

20. Secondary Outcome: Standardized Morning Erections Question (SMEQ) Score at Month 9
Description: as for outcome 19
Time Frame: Month 9
Population: All randomized participants who received at least 1 dose of study drug and had SMEQ measurement at Month 9.
Measure: Number; unit: participants
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 114 | 122 | 115
participants
  Yes, regularly | 7 | 9 | 7
  Less frequently than in the past | 21 | 19 | 9
  Only occasionally | 36 | 26 | 27
  Never | 39 | 61 | 65
  Missing | 11 | 7 | 7

21. Secondary Outcome: Standardized Morning Erections Question (SMEQ) Score at Month 13.5
Description: as for outcome 19
Time Frame: Month 13.5
Population: All randomized participants who received at least 1 dose of study drug and had SMEQ measurement at Month 13.5.
Measure: Number; unit: participants
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 100 | 114 | 106
participants
  Yes, regularly | 13 | 15 | 13
  Less frequently than in the past | 22 | 24 | 18
  Only occasionally | 31 | 30 | 27
  Never | 32 | 40 | 42
  Missing | 2 | 5 | 6

22. Secondary Outcome: Change From Baseline in 26-item Expanded Prostate Cancer Index Composite (EPIC-26) Questionnaire Score
Description: EPIC-26 (participants) contains 26 items and 5 domains: Urinary Incontinence (Items 1-4), Urinary Irritative/Obstructive (Items 5-8), Bowel (Items 10-15), Sexual (Items 16-21), and Hormonal (Items 22-26). Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0 to 100 scale for each domain, with higher scores representing better health-related quality of life. Responses are based on experiences during the previous 4 weeks. The Mixed Model for Repeated Measures (MMRM) analysis was used to calculate Least Squares (LS) mean and 95% confidence interval (CI). LS mean values are adjusted for baseline domain score, treatment, country, visit, visit-by-treatment, age group, and age group-by-treatment (if significant at p<0.10).
Time Frame: Randomization (Baseline), Months 9 and 13.5
Population: All randomized participants who received at least 1 dose of study drug, had baseline and at least 1 post-baseline EPIC-26 scores measurement at Month 9 and Month 13.5.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 139 | 142 | 141
units on a scale
  Urinary Incontinence - Month 9 | 34.08 [29.31 to 38.86] | 31.12 [26.74 to 35.51] | 30.59 [25.85 to 35.33]
  Urinary Incontinence - Month 13.5 | 37.41 [32.56 to 42.26] | 35.54 [31.10 to 39.97] | 35.44 [30.65 to 40.23]
  Urinary Irritative/Obstructive - Month 9 | 13.83 [11.54 to 16.12] | 13.28 [11.19 to 15.37] | 12.26 [10.01 to 14.51]
  Urinary Irritative/Obstructive - Month 13.5 | 13.86 [11.53 to 16.20] | 13.82 [11.70 to 15.94] | 12.30 [0.01 to 14.60]
  Bowel - Month 9 | 5.94 [3.71 to 8.17] | 6.27 [4.22 to 8.33] | 6.48 [4.31 to 8.65]
  Bowel - Month 13.5 | 6.87 [4.67 to 9.08] | 6.49 [4.46 to 8.52] | 6.78 [4.61 to 8.94]
  Sexual - Month 9 | 27.53 [21.64 to 33.42] | 20.66 [15.27 to 26.06] | 17.98 [12.14 to 23.81]
  Sexual - Month 13.5 | 36.55 [30.03 to 43.06] | 32.58 [26.60 to 38.56] | 33.37 [26.95 to 39.79]
  Hormonal - Month 9 | 1.72 [-0.81 to 4.26] | 2.72 [0.36 to 5.08] | -0.18 [-2.67 to 2.31]
  Hormonal - Month 13.5 | 2.48 [0.10 to 4.87] | 2.92 [0.76 to 5.08] | 3.01 [0.67 to 5.36]
Statistical Analysis 1: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.196, Mixed Models Analysis — P-value is for Urinary Incontinence - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 3.49, 95% CI 2-sided [-1.82 to 8.80], Standard Error of Mean 2.70
Statistical Analysis 2: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.841, Mixed Models Analysis — P-value is for Urinary Incontinence - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.53, 95% CI 2-sided [-4.69 to 5.75], Standard Error of Mean 2.65
Statistical Analysis 3: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.474, Mixed Models Analysis — P-value is for Urinary Incontinence - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 1.98, 95% CI 2-sided [-3.45 to 7.40], Standard Error of Mean 2.76
Statistical Analysis 4: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.971, Mixed Models Analysis — P-value is for Urinary Incontinence - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.10, 95% CI 2-sided [-5.21 to 5.41], Standard Error of Mean 2.70
Statistical Analysis 5: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.236, Mixed Models Analysis — P-value is for Urinary Irritative/Obstructive - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 1.57, 95% CI 2-sided [-1.03 to 4.17], Standard Error of Mean 1.32
Statistical Analysis 6: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.429, Mixed Models Analysis — P-value is for Urinary Irritative/Obstructive - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 1.02, 95% CI 2-sided [-1.52 to 3.56], Standard Error of Mean 1.29
Statistical Analysis 7: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.252, Mixed Models Analysis — P-value is for Urinary Irritative/Obstructive - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 1.56, 95% CI 2-sided [-1.12 to 4.24], Standard Error of Mean 1.36
Statistical Analysis 8: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.251, Mixed Models Analysis — P-value is for Urinary Irritative/Obstructive - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 1.52, 95% CI 2-sided [-1.08 to 4.11], Standard Error of Mean 1.32
Statistical Analysis 9: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.671, Mixed Models Analysis — P-value is for Bowel - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = -0.54, 95% CI 2-sided [-3.03 to 1.95], Standard Error of Mean 1.27
Statistical Analysis 10: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.868, Mixed Models Analysis — P-value is for Bowel - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = -0.21, 95% CI 2-sided [-2.64 to 2.23], Standard Error of Mean 1.24
Statistical Analysis 11: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.938, Mixed Models Analysis — P-value is for Bowel - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 0.10, 95% CI 2-sided [-2.37 to 2.57], Standard Error of Mean 1.25
Statistical Analysis 12: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.813, Mixed Models Analysis — P-value is for Bowel - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = -0.29, 95% CI 2-sided [-2.69 to 2.12], Standard Error of Mean 1.22
Statistical Analysis 13: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis — P-value is for Sexual - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 9.55, 95% CI 2-sided [3.10 to 15.99], Standard Error of Mean 3.28
Statistical Analysis 14: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.403, Mixed Models Analysis — P-value is for Sexual - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 2.69, 95% CI 2-sided [-3.63 to 9.00], Standard Error of Mean 3.21
Statistical Analysis 15: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.406, Mixed Models Analysis — P-value is for Sexual - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 3.18, 95% CI 2-sided [-4.34 to 10.69], Standard Error of Mean 3.82
Statistical Analysis 16: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.832, Mixed Models Analysis — P-value is for Sexual - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = -0.79, 95% CI 2-sided [-8.11 to 6.53], Standard Error of Mean 3.72
Statistical Analysis 17: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.197, Mixed Models Analysis — P-value is for Hormonal - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 1.90, 95% CI 2-sided [-0.99 to 4.79], Standard Error of Mean 1.47
Statistical Analysis 18: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.045, Mixed Models Analysis — P-value is for Hormonal - Month 9; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = 2.89, 95% CI 2-sided [0.06 to 5.72], Standard Error of Mean 1.44
Statistical Analysis 19: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.692, Mixed Models Analysis — P-value is for Hormonal - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = -0.53, 95% CI 2-sided [-3.16 to 2.10], Standard Error of Mean 1.34
Statistical Analysis 20: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.943, Mixed Models Analysis — P-value is for Hormonal - Month 13.5; [statistical method as in outcome 3, analysis 1]; LS Mean Differences = -0.09, 95% CI 2-sided [-2.65 to 2.46], Standard Error of Mean 1.30

23. Secondary Outcome: Change in Penile Length and Girth
Description: Measurements were performed with the penis in the flaccid state. The stretched penile length was measured from the tip of the glans to the pubopenile skin junction while applying tension to maximally stretch the penis. The penile circumference at midshaft was measured. All measurements were taken with a paper ruler to the nearest 0.5 centimeter (cm). The analysis of covariance (ANCOVA) was used to calculate Least Square (LS) mean and 95% confidence interval (CI). LS mean values are adjusted for treatment, baseline, age group and country.
Time Frame: Randomization (Baseline), Month 9
Population: All randomized participants who received at least 1 dose of study drug and had penile measurements at Baseline and Month 9.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeter (mm)
Arm/Group | Tadalafil 5 mg OaD | Tadalafil 20 mg PRN | Placebo
Number analyzed (Participants) | 139 | 142 | 141
millimeter (mm)
  Length | -1.53 [-5.54 to 2.47] | -7.26 [-11.04 to -3.49] | -5.73 [-9.68 to -1.78]
  Girth | 0.03 [-3.09 to 3.15] | 0.82 [-2.11 to 3.75] | -2.34 [-5.43 to 0.75]
Statistical Analysis 1: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.028, ANCOVA — P-value is for length; ANCOVA model included terms for treatment, baseline, age group and country; LS Mean Differences = 4.20, 95% CI 2-sided [0.47 to 7.93], Standard Error of Mean 1.89
Statistical Analysis 2: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.413, ANCOVA — P-value is for length; ANCOVA model included terms for treatment, baseline, age group and country; LS Mean Differences = -1.53, 95% CI 2-sided [-5.20 to 2.14], Standard Error of Mean 1.87
Statistical Analysis 3: Comparison: Tadalafil 5 mg OaD vs Placebo; Test type: Superiority or Other; p = 0.112, ANCOVA — P-value is for girth; ANCOVA model included terms for treatment, baseline, age group and country; LS Mean Differences = 2.37, 95% CI 2-sided [-0.55 to 5.30], Standard Error of Mean 1.49
Statistical Analysis 4: Comparison: Tadalafil 20 mg PRN vs Placebo; Test type: Superiority or Other; p = 0.031, ANCOVA — P-value is for girth; ANCOVA model included terms for treatment, baseline, age group and country; LS Mean Differences = 3.16, 95% CI 2-sided [0.29 to 6.03], Standard Error of Mean 1.46

ADVERSE EVENTS:
Groups:
- Screen - BNSRP: Had bilateral nerve-sparing radical prostatectomy (BNSRP) surgery during Screening Period.
- Tadalafil 5 mg OaD (Double-Blind Period/Washout Period): Tadalafil 5 mg once a day (OaD) + Placebo as required/on demand (PRN) for 9 months during Double-Blind, Placebo-Controlled Treatment Period, followed by a 6-week, Drug-Free Washout Period.
- Tadalafil 20 mg PRN (Double-Blind Period/Washout Period): Placebo OaD + Tadalafil 20 mg PRN for 9 months during Double-Blind, Placebo-Controlled Treatment Period, followed by a 6-week, Drug-Free Washout Period.
- Placebo (Double-Blind Period/Washout Period): Placebo OaD + Placebo PRN for 9 months during Double-Blind, Placebo-Controlled Treatment Period, followed by a 6-week, Drug-Free Washout Period.
- Tadalafil 5 mg OaD (Open-Label Period): Tadalafil 5 mg OaD + Placebo PRN for 9 months during Double-Blind, Placebo-Controlled Treatment Period, followed by a 6-week, Drug-Free Washout Period, and a 3-month, Open-Label Period with tadalafil 5 mg OaD.
- Tadalfil 20 mg PRN (Open-Label Period): Placebo OaD + Tadalafil 20 mg PRN for 9 months during Double-Blind, Placebo-Controlled Treatment Period, followed by a 6-week, Drug-Free Washout Period, and a 3-month, Open-Label Period with tadalafil 5 mg OaD.
- Placebo (Open-Label Period): Placebo OaD + Placebo PRN for 9 months during Double-Blind, Placebo-Controlled Treatment Period, followed by a 6-week, Drug-Free Washout Period, and a 3-month, Open-Label Period with tadalafil 5 mg OaD.
Arm/Group | Screen - BNSRP | Tadalafil 5 mg OaD (Double-Blind Period/Washout Period) | Tadalafil 20 mg PRN (Double-Blind Period/Washout Period) | Placebo (Double-Blind Period/Washout Period) | Tadalafil 5 mg OaD (Open-Label Period) | Tadalfil 20 mg PRN (Open-Label Period) | Placebo (Open-Label Period)
Serious Adverse Events (participants affected / at risk) | 6/583 | 2/139 | 3/143 | 10/141 | 1/139 | 1/143 | 2/141
Other Adverse Events (participants affected / at risk) | 114/583 | 50/139 | 52/143 | 40/141 | 11/139 | 18/143 | 9/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Screen - BNSRP (N=583) | Tadalafil 5 mg OaD (Double-Blind Period/Washout Period) (N=139) | Tadalafil 20 mg PRN (Double-Blind Period/Washout Period) (N=143) | Placebo (Double-Blind Period/Washout Period) (N=141) | Tadalafil 5 mg OaD (Open-Label Period) (N=139) | Tadalfil 20 mg PRN (Open-Label Period) (N=143) | Placebo (Open-Label Period) (N=141)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Event resulted in death
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hernia obstructive (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine flow decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocele (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Screen - BNSRP (N=583) | Tadalafil 5 mg OaD (Double-Blind Period/Washout Period) (N=139) | Tadalafil 20 mg PRN (Double-Blind Period/Washout Period) (N=143) | Placebo (Double-Blind Period/Washout Period) (N=141) | Tadalafil 5 mg OaD (Open-Label Period) (N=139) | Tadalfil 20 mg PRN (Open-Label Period) (N=143) | Placebo (Open-Label Period) (N=141)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Androgen deficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoprolactinaemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Posterior capsule opacification (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bowel movement irregularity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (8) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 5 (6) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue geographic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Local swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 2 (2)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 5 (5) | 5 (5) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 21 (23) | 3 (4) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anastomotic complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 7 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incision site blister (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incision site complication (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Open wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 13 (14) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Testicular injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthroscopy (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood luteinising hormone decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood selenium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood selenium increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood testosterone decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oestradiol increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine output increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 5 (5) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (7) | 5 (7) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Essential tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 9 (10) | 5 (11) | 11 (16) | 6 (7) | 1 (2) | 2 (2) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orgasm abnormal (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder irritation (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder tamponade (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urge incontinence (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 34 (34) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile curvature (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scar pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthroscopic surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder catheterisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Circumcision (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental implantation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Knee operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polypectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wart excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocele (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days